CLINICAL TRIAL: NCT06108648
Title: Efficacy of Lavender Essential Oil Chest Wraps in Improving Cough and Respiratory Distress in Infants With Bronchiolitis: a Multicenter Randomized Controlled Trial
Brief Title: Efficacy of Lavender Essential Oil Chest Wraps in Infants With Bronchiolitis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Fabiola Stollar, Attending Physician, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-01116
Record Dates: First submitted 2023-10-08; First posted 2023-10-31 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Bronchiolitis
Keywords: bronchiolitis; infant; cough; essential oil; lavendula; complementary therapies
MeSH Terms: conditions — Bronchiolitis; Cough | interventions — lavender oil; Olive Oil

STUDY DESIGN:
Intervention Model Description: Patients are randomized to receive standard care with additional lavender essential oil chest wrap during two nights of hospitalization or standard care alone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lavender oil (Experimental): Lavender chest wrap:
  Before the first application pour 10-15 ml of lavender essential oil 10% evenly on the cotton cloth. Put the soaked cotton in the plastic bag, close it and put it to heat in two heating pads (2-5 minutes) so that the oil is distributed on all the fabric. Place the cotton cloth around the patient's chest. Cover the cotton cloth with a woolen fabric that is 2 cm larger than the cotton cloth.
  Interventions: Drug: Lavender essential oil 10%, diluted in 90% olive oil
- Control (Active Comparator): Standard care: supportive measures according to national standards.
  Interventions: Other: Control

INTERVENTIONS:
Drug: Lavender essential oil 10%, diluted in 90% olive oil — Lavender chest wrap:
  Before the first application pour 10-15 ml of lavender essential oil 10% evenly on the cotton cloth.
  Put the soaked cotton in the plastic bag, close it and put it to heat in two heating pads (2-5 minutes) so that the oil is distributed on all the fabric. Place the cotton cloth around the patient's chest.
  Cover the cotton cloth with a woolen fabric that is 2 cm larger than the cotton cloth.
  Arms: Lavender oil
Other: Control — Standard care according to national standards.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to learn if lavender essential oil chest wraps relieve cough in infants with bronchiolitis compared to standard care. Furthermore, the researchers will evaluate if breathing difficulties, nighttime awakening and impact on parents will be improved by the lavender oil chest wraps. Infants will be randomized to receive standard care with the addition of lavender oil chest wraps or to receive standard care alone. The study will take place in two locations in Switzerland, at the Geneva University Hospital and the Fribourg Cantonal Hospital.

ELIGIBILITY:
Inclusion criteria:

* Bronchiolitis: clinical diagnosis based on the combination of respiratory distress (tachypnea, grunting, nasal flaring, retractions, and/or need for supplementary oxygen) and fine crackles sometimes accompanied by wheezing on auscultation.
* Hospitalization.
* Written informed consent.

Exclusion criteria:

* Patients with underlying diseases that impact respiratory or heart function (congenital heart disease, congenital malformation of the lung or airway system and severe chronic lung disease).
* More than 3 episodes of bronchiolitis.
* Critically ill infants who have an immediate need for intensive care unit (ICU) admission.
* Respiratory deterioration needing Continuous positive airway pressure (CPAP) or transfer to ICU during study enrollment.
* Atopic dermatitis, eczema or other skin lesions (particularly on the chest).
* Oncologic disease.
* Premature infants with mild bronchopulmonary dysplasia will not be excluded.

Max Age: 11 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Cough frequency | Up to 2 days
  Number of coughs per hour measured with Hyfe CoughMonitor (Hyfe Inc)

SECONDARY OUTCOMES:
Crying episodes | Up to 2 days
  Number of crying episodes noted by parents on crying calendar
Respiratory rate | Baseline, 1 hour, 4 hours
  Number of breaths per minute
Oxygen supplementation requirement | Immediately at discharge from hospital
  Presence of oxygen supplementation during hospital stay (yes/no)
Oxygen supplementation duration | Immediately at discharge from hospital
  Number of hours of oxygen supplementation
Maximum oxygen supplementation | Immediately at discharge from hospital
  Maximum oxygen flow in L/min
Hospital length of stay | Immediately at discharge from hospital
  Hospital length of stay in number of days, Geneva site only
Parental satisfaction assessed with patient satisfaction questionnaire | Immediately at discharge from hospital
  Satisfaction of parents will be measured by a 10-item, four-point Likert scale questionnaire that has a 3-dimensional structure, i.e. overall satisfaction; perceived effectiveness; parental information and involvement. Scale range from 1 (not at all) to 4 (a lot). Higher scores indicate greater satisfaction.
Impact on parents assessed by the "Impact of Bronchiolitis Hospitalization Questionnaire" (IBHQ) | Immediately at discharge from hospital
  Impact from the hospitalization on parents will be measured using IBHQ, a 46-item, four-point Likert scale that has a 12-dimensional structure, i.e. worries and distress; fear for future; guilt; impact on daily organization; physical impact; impact on behaviour with hospitalized child; financial impact; disturbed breastfeeding; physical reaction of hospitalized child; impact on feeding of hospitalized child; impact on behaviour with other children; sibling's reaction. Scale ranges from 1 (not at all) to 4 (a lot). Higher scores indicate higher impact on parents.

CONTACTS AND LOCATIONS:
Overall Officials: Klara Posfay-Barbe, MD, PhD, Study Director — Children's' Hospital, University Hospital of Geneva, Switzerland
Locations (2):
- Switzerland (2):
  - Clinique de pediatrie, HFR Fribourg - Hopital cantonal, Switzerland, Fribourg
  - Children's' Hospital, University Hospital of Geneva, Switzerland, Geneva

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board, Independent Ethics Committee, or Research Ethics Board, as applicable, and executes a data use/sharing agreement with the Geneva University Hospitals HUG.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigator who has approval from an Institutional Review Board, Independent Ethics Committee, or Research Ethics Board, as applicable, and executes a data use/sharing agreement with the Geneva University Hospitals HUG.
URL: https://recherche.hug.ch/